CLINICAL TRIAL: NCT02964143
Title: Prospective, Randomized, Controlled Clinical Investigation to Compare the Safety and Performance of a Combination of Autologous Platelet-rich Plasma (PRP) and Hyaluronic Acid Prepared With Cellular MatrixTM to Those of Ostenil® Plus and to Those of PRP Alone in the Treatment of Mild to Moderate Osteoarthritis of the Knee
Brief Title: Clinical Investigation to Compare the Safety and Efficacy of Cellular Matrix to Those of Ostenil® Plus and to Those of PRP Only
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-OA-001
Record Dates: First submitted 2016-10-13; First posted 2016-11-15 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All patients will undergo blood collection, whatever treatment they will receive. The day of each treatment session, a specially trained staff member, who won't be otherwise related to the study, will perform blood withdrawal and prepare the treatment according to the randomization code in a separate -but neighboring- room. This staff member will then deliver the treatment to the ward where the clinician will inject it into the patient's knee. To preserve patient's blindness, a screen will be placed in order to prevent him/her from seeing the whole procedure (from blood withdrawal to treatment injection).
  Evaluation of primary and secondary endpoints will be performed by a blinded assessor who will not know which treatment (PRP/HA combination, HA alone, or PRP alone) was given to the patient. The blinded assessor will not perform any other study-related procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Patients from this group will be treated with a combination of platelet-rich plasma (PRP) and hyaluronic acid (HA) prepared with the Cellular Matrix / A-CP HA medical device
  Interventions: Device: Cellular Matrix / A-CP HA
- Control group 1 (Active Comparator): Patients from this group will be treated with a well-recognized hyaluronic acid named Ostenil® Plus
  Interventions: Device: Ostenil® Plus
- Control group 2 (Active Comparator): Patients from this group will be treated with PRP alone, prepared with RegenKit-BCT-1
  Interventions: Device: RegenKit-BCT-1

INTERVENTIONS:
Device: Cellular Matrix / A-CP HA — Treatment with 2 injections of Cellular Matrix / A-CP HA Kit, administered 2 months apart; Cellular Matrix / A-CP HA Kit is designed for the safe, rapid and extemporaneous preparation of a cellular matrix of autologous PRP combined with HA. The Cellular Matrix / A-CP HA Kit is a single-use medical device including hematology tubes (A-CP HA tube), designed for blood collection and PRP/HA preparation after 5 min centrifugation. This tube contains a non-crosslinked hyaluronic acid (MW 1550 kDa) solution, a gel acting as a cell separator, and a sodium citrate acting as an anticoagulant. During centrifugation, the separator gel moves to form a barrier that separates red blood cells from other blood components. The HA, which migrates to the top of the gradient during centrifugation, can be mixed with PRP in order to give rise to a ready-to-use PRP/HA preparation.
  Arms: Experimental group
Device: Ostenil® Plus — Treatment with 2 injections of Ostenil® Plus, administered one week apart; Ostenil® Plus is a solution of sodium hyaluronate obtained by fermentation, containing 0.5% mannitol, a free radical scavenger, which helps to stabilize the chains of sodium hyaluronate. The product is intended to be used for pain and restricted mobility in degenerative and traumatic changes of the knee joint.
  Arms: Control group 1
Device: RegenKit-BCT-1 — Treatment with 2 injections of RegenKit-BCT-1, administered 1 month apart; RegenKit-BCT-1 is designed for the safe, rapid and extemporaneous preparation of autologous platelet-rich plasma. RegenKit-BCT-1 is a single-use medical device including an hematology tube (Regen BCT tube), designed for blood collection and PRP preparation after 5 min centrifugation, and all necessary material for venipuncture and PRP injection. The Regen BCT tube contains a gel acting as a cell separator and a sodium citrate acting as an anticoagulant. During centrifugation, the separator gel moves to form a barrier that separates red blood cells from other blood components.
  Arms: Control group 2

SUMMARY:
Platelet-rich plasma (PRP) is an autologous product prepared from the patient's own blood, representing a powerful source of platelet-derived growth factors, particularly useful in the field of regenerative medicine. The active and sequential secretion of these growth factors induces different cell signaling cascades that activate angiogenesis, cell proliferation, cell differentiation, eventually leading to new matrix synthesis and tissue regeneration.

The potential benefits from the use of PRP for the treatment of cartilage defects rely on a number of studies conducted in validated animal models or in vitro, demonstrating the ability of PRP to stimulate collagen production and proteoglycans synthesis, as well as the proliferation and differentiation of mesenchymal stem cells into chondrocytes. Additionally, an increasing number of clinical studies shows an improvement of symptoms, most especially pain, without any occurrence of serious adverse events.

Hyaluronic acid (HA), as one of the major components of the synovial fluid surrounding the cartilage, assumes an important role in the viscoelastic properties of the articular cartilage, conferring its shock absorbing and lubricating functions.

It was demonstrated that rheological properties of synovial fluid decrease with aging and in patients suffering from osteoarthritis. Nowadays, intra-articular injections of hyaluronic acid represent a well recommended therapeutic option to relieve osteoarthritic symptoms, conferring a mechanical action on joints structures, thus leading to reduced pain and improved joint function Based on these data, it seems reasonable to hypothesize that a combination of both PRP and hyaluronic acid could provide greater benefits compared to the administration of each product alone, as their effects on osteoarthritis improvement are based on different mechanisms of action. In fact, on one side PRP promotes cartilage regeneration, while on the other side the HA acts as 3-dimensional support mesh for PRP, providing optimal release of platelets growth factors, strengthening and extending in time the activity of PRP.

Cellular MatrixTM is a CE-marked class III medical device manufactured by the Swiss company RegenLab SA. Cellular MatrixTM allows to prepare autologous PRP combined with a non-crosslinked hyaluronic acid in a safe, rapid manner and in a single step. The PRP/HA combination is intended to be injected intra-articularly, in order to relieve osteoarthritic symptoms and to improve joint mobility and function. Therefore, the PRP/HA combination might represent a novel therapeutic option for patient suffering from knee osteoarthritis.

This study will evaluate whether the effects of a PRP/HA combination prepared with Cellular Matrix™, when injected intra-articularly for the treatment of mild to moderate knee osteoarthritis, are superior to those of a well-recognized hyaluronic acid treatment (Ostenil® Plus), on one hand, and to those of PRP alone, on the other hand.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee osteoarthritis of a unilateral knee, characterized by pain at walking (WOMAC A1 score assessed over the previous 24 hours on a 100-mm VAS: 50 ≤ WOMAC A1 ≤ 90) or reduced joint function (total WOMAC C score assessed or over the previous 24 hours on a 100-mmVAS: 50 ≤ WOMAC A1 ≤ 90)
* Femoro-tibial knee osteoarthritis defined according to ACR criteria
* Bilateral knee osteoarthritis is allowed, provided the contralateral knee is characterized by a maximum pain of 30 on a 0 to 100 mm scale and doesn't require systemic analgesic treatment, with the exception of paracetamol up to the maximum dose of 4 g per day
* Radiographic femoro-tibial knee osteoarthritis (radiograph not older than 3 months) Kellgren & Lawrence grades of II-III
* Outpatient capable of walking 50 meters without assistance
* Signature of the informed consent form
* Capable of understanding the study's imperatives, as well as written instructions
* Capable of filling-out evaluation questionnaires

Exclusion Criteria:

* Radiographic femoro-tibial knee osteoarthritis Kellgren & Lawrence grades of I or IV
* Bilateral knee osteoarthritis, characterized by pain greater than 30 of both knees evaluated on a 0 to 100-mm scale and requiring systemic analgesic treatment or paracetamol greater than 4g/ day
* Viscosupplementation in the past 3 months
* Corticosteroid injection in the past 3 months
* PRP or PRP/HA injection in the past 12 months
* Any surgery of the knee planned during the next 6 months
* Systematic use of corticosteroids (except those that are inhaled) or level III analgesics in the past 3 months and NSAID during the past month
* Treatment with slow-acting anti-rheumatic drugs (diacerhein, soybean or avocado unsaponifiables, chondroitin sulfate, glucosamine) started in the past 6 months
* History of allergy to hyaluronic acid
* Auto-immune disease (rheumatoid arthritis, lupus)
* Surgery of the affected knee in the past 3 months
* Infection of the affected knee in the past 6 months
* Rheumatologic disorder other than arthritis
* Clinical evidence of local inflammation such as redness or heat of the joint
* Any knee surgery planned within 6 months
* Hereditary or acquired hematologic or clotting disorders, such as drepanocytosis, platelet dysfunction, thrombocytopenia (<150'000 platelets/mm3), etc.
* Anemia (Hemoglobin < 10g/dl)
* Anticoagulant treatment (patients under antiaggregant treatment can take part to this study as long as their clotting time (CT) is within the reference value)
* Acute infection
* Malignant disease (especially bone and hematological)
* Recent fever or serious disorders (cardiovascular pathology, active gastroduodenal ulcer, digestive hemorrhage, liver disease, etc.)
* Patient with renal impairment (creatinine clearance below 45 ml / min)
* Patient with liver failure, pending or who have recently received a liver transplant
* Infectious diseases
* Pregnancy or breastfeeding or planning pregnancy during the course of the study
* Immunosuppression
* Insulin-dependent diabetic patient
* Participation ongoing or in the past 3 months in another clinical study
* Participation to another osteoarthritis clinical study during the past year
* Refusal to sign or inability to give Informed Consent
* Patient unable to submit to the constraints of the protocol, including patient whose mental condition does not allow him to understand the nature, objectives and possible consequences of the study
* Any other reason which, in the opinion of the investigator, may interfere with the proper conduct of the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Variation of the pain between baseline and Month 6 | 6 months
  For each group, pain will be evaluated using the WOMAC A subscale; each item of this subscale will be scored using a 100-mm VAS (Visual Analogue Scale) at baseline and Month 6. The total WOMAC A score will be reported as a summed score of this subscale.

SECONDARY OUTCOMES:
Variation of pain between baseline and Month 1, Month 2 and Month 4 | 1, 2 and 4 months
  For each group, pain will be evaluated using the WOMAC A subscale; each item of this subscale will be scored using a 100-mm VAS (Visual Analogue Scale) at baseline, Month 1, Month 2, and Month 4. The total WOMAC A score will be reported as a summed score of all items of this subscale.
Variation of stiffness between baseline and Month 1, Month 2, Month 4 and Month 6 | 1, 2, 4 and 6 months
  For each group, stiffness will be evaluated using the WOMAC B subscale; each item of this subscale will be scored using a 100-mm VAS (Visual Analogue Scale) at baseline, Month 1, Month 2, Month 4 and Month 6. The total WOMAC B score will be reported as a summed score of all items of this subscale.
Variation of physical function between baseline and Month 1, Month 2, Month 4 and Month 6 | 1, 2, 4 and 6 months
  For each group, physical function will be evaluated using the WOMAC C subscale; each item of this subscale will be scored using a 100-mm VAS (Visual Analogue Scale) at baseline, Month 1, Month 2, Month 4 and Month 6. The total WOMAC C score will be reported as a summed score of all items of this subscale.
Variation of overall knee osteoarthritis symptoms between baseline and Month 1, Month 2, Month 4 and Month 6 | 1, 2, 4 and 6 months
  For each group, overall knee osteoarthritis will be evaluated using the total WOMAC questionnaire; each item of this questionnaire will be scored using a 100-mm VAS (Visual Analogue Scale) at baseline, Month 1, Month 2, Month 4 and Month 6. The total WOMAC score will be reported as a summed score of all items of the questionnaire.
Variation of the quality of life between baseline and all time points | 1, 2, 4 and 6 months
  Quality of life will be assessed using the SF-36 questionnaire that will be given to patients at each visit throughout the study.
Patient Global Assessment of the treatment received | 6 months
Clinician Global Assessment of the treatment | 6 months
Percentage of OMERACT-OARSI responders at Month 1, Month 2, Month 4 and Month 6 | 1, 2, 4 and 6 months
Percentage of patients requiring an injection of the combination of PRP/HA prepared with Cellular Matrix / A-CP HA at Month 6 | 6 months
Number of local and systemic side effects throughout the study period | 12 months
Cartilage structure | 6 and 12 Months
  The cartilage structure will be evaluated on the basis of Magnetic Resonance Imaging (MRI) assays at baseline (before receiving the treatment), 6 and 12 months. Differences on the T1 relaxation time parameter will be evaluated at different time points.

IPD SHARING:
Plan to Share IPD: No